CLINICAL TRIAL: NCT06732674
Title: A 54-week, Multi-centre, 2-arm, Randomised Controlled Trial to Assess Home Monitoring for Lung Function and Patient Reported Outcome Measurements Vs. Usual Care in RheuMatic Disease-associated Interstitial Lung Disease: the RMD-mILDer Trial
Brief Title: Home Based Clinical Management of Interstitial Lung Disease in Systemic Rheumatic Diseases
Acronym: RMD-mILDer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, Anna-Maria Hoffmann-Vold, Prof Dr med, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 535561
Record Dates: First submitted 2024-12-02; First posted 2024-12-13 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Interstitial Lung Disease with Progressive Fibrotic Phenotype in Diseases Classified Elsewhere; Systemic Sclerosis Pulmonary; Dermatomyositis; Rheumatoid Arthritis; Sjogren Syndrome with Lung Involvement; Connective Tissue Diseases
Keywords: home monitoring; remote monitoring; interstitial lung disease; rheumatic disease; lung fibrosis; Systemic sclerosis; Dermatomyositis; Sjøgren
MeSH Terms: conditions — Dermatomyositis; Arthritis, Rheumatoid; Connective Tissue Diseases; Lung Diseases, Interstitial; Rheumatic Diseases; Pulmonary Fibrosis; Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: international, multi-center, 2-arm, 54-week, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Scheduled hospital visits every 6 months
- Home monitoring (Experimental): Home monitoring strategy with remote patient data observation twice a week
  Interventions: Diagnostic Test: A home monitoring strategy with event driven management

INTERVENTIONS:
Diagnostic Test: A home monitoring strategy with event driven management — Bi-weekly home monitoring with forced vital capacity (FVC), patient reported outcome measures (PROMs), at-home measures of blood oxygen levels (SpO2) during 1-minute-sit-to-stand test (1MSTS) and temperature with algorithm based risk evaluation of deterioration and infection and consecutive event driven management
  Arms: Home monitoring

SUMMARY:
The RMD-mILDer trial is a home monitoring strategy trial aiming to improve management of interstitial lung disease related to rheumatic diseases applying eHealth technology.

It is planned as a 2 arm 54 week multi-centre randomised controlled trial to assess outcome of home monitoring with bi-weekly serial forced vital capacity- and patient reported outcome-measurements compared to standard of care with fixed-interval hospital visits in adult patients with rheumatic disease associated interstitial lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* Systemic rheumatic disease (Systemic sclerosis (SSc), rheumatoid arthritis (RA), idiopathic inflammatory myopathies including antisynthetasis syndromes (IIM), mixed connective tissue disease (MCTD) or Sjøgrens disease (SjD)) classifiable by disease-specific classification criteria
* Diagnosed interstitial lung disease (ILD) on high resolution computed tomography (HRCT) ≥ 1 year prior to randomization, not explained by other diseases or exposures
* On stable standard of care treatment 6 months prior to randomization
* Participants must be able to understand and follow trial procedures including completion of questionnaires regarding Patient Reported Outcome measures
* Participants must have access to the internet, and experience in using smartphones or other electronic devices with internet access
* Signed informed consent form

Exclusion Criteria:

* Severe heart failure with ejection fraction (EF) < 30%
* Chronic renal failure G4 or more (defined by KDIGO) with glomerular filtration rate (eGFR) < 30 mL/min using Cockroft-Gault formula.
* End stage lung disease with forced vital capacity (FVC) < 50% and/or diffusion capacity for carbon monoxide (DLCO) < 40% or coexisting severe other lung diseases (e.g. chronic obstructive pulmonary disease, emphysema)
* Airway obstruction (pre-bronchodilator FEV1/FVC < 0.7) (FEV1 is defined as forced expiratory volume in 1 sec)
* In the opinion of the investigator, other clinically significant pulmonary abnormalities
* Significant pulmonary hypertension defined by the following: Previous clinical or echocardiographic evidence of significant right heart failure OR history of right heart catheterization showing a cardiac index </= 2 L/min/m2 OR pulmonary hypertension requiring therapy with epoprostenol/treprostinil
* Active treatment for cancer or non-curable cancer
* Relative contraindications to performing spirometry, as specified in ATS/ERS guidelines.
* Ongoing Prednisolone ≥ 20 mg/day at inclusion
* Unable to speak, write and read Norwegian, German or Romanian in the respective country of inclusion.
* Unable to perform good quality measurements of FVC on the home-device comparable to results on an in-hospital device, after training.
* Pregnancy or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Assess whether home monitoring identifies disease progression earlier than monitoring by fixed-interval hospital visits. | 54 weeks
  Time from baseline to disease progression assessed as first forced vital capacity (FVC) ≥5% decline (assessed by hospital FVC measurements) or non-elective hospitalization due to respiratory cause.

SECONDARY OUTCOMES:
Estimate effects of home monitoring compared to fixed-interval hospital visits on change in FVC | after 54 weeks
  Absolute change from baseline in FVC (mL) and absolute change from baseline in FVC (% predicted).
Estimate effects of home monitoring compared to fixed-interval hospital visits on FVC decline >10% events. | baseline to week 54
  Proportion of patients who experience at least one FVC decline >= 10% event from baseline
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported respiratory symptoms | baseline to week 54
  Change in "Living with pulmonary fibrosis score" (LPF) total score, as well as the subdomains physical health, emotional well-being, social impact, functionality and daily activities as well as cognitive function where lower values indicate quality of life
Estimate effects of home monitoring compared to fixed hospital visits on progressive pulmonary fibrosis events. | baseline to week 54
  Proportion of patients who experience a progressive pulmonary fibrosis event defined as fibrosing ILD fulfilling ≥2 (out of 3) criteria (worsening respiratory symptoms, radiological progression, and physiological progression (absolute decline in FVC ≥ 5% predicted within 1 year follow up OR absolute decline in diffusion capacity for carbon monoxide (DLCO) ≥10% predicted within 1 year of follow up) occurring within the past year with no alternative explanation in a patient with ILD.

OTHER OUTCOMES:
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported symptoms related to the rheumatic disease (RMD) | baseline to week 54
  Change in visual analogue scale (VAS) on RMD from 0 - 10 with higher values indicating more symptoms
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported general well-being | baseline to week 54
  Change in VAS on the patients global health from 0 - 10 with higher values indicating more symptoms
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported health related quality of life | baseline to week 54
  Change in the EuroQol Eq-5D-5L questionnaire with the following domains: Mobility, self-care, usual activities, pain/discomfort, anxiety/depression. The score typically ranges from 0 (representing a health state equivalent to death) to 1 (representing perfect health).
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported disability to perform daily tasks and carry out basic activity | baseline to week 54
  Change in Health Assessment Questionaire (HAQ) covering eight different domains: Dressing and grooming, arising, eating, walking, hygiene, reach, gripping and activities.
  The HAQ has 20 questions. The score reaches from 0 (no incapacity) to 3 (full incapacity)
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported pain, fatigue and dryness in included patients with interstitial lung disease (ILD) related to Sjøgrens disease (SjD-ILD) | baseline to week 54
  Change in EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) with a range of 0 - 10, with higher values indicating more symptoms.
Estimate effects of home monitoring compared to fixed-interval hospital visits on the patient reported impact of the diseases in included patients with ILD related to systemic sclerosis | baseline to week 54
  Change in EULAR Systemic Sclerosis Impact of Disease (ScleroID) questionnaire whereby higher counts on a scale from 0-100 would indicate more impact
Estimate effects of home monitoring compared to fixed-interval hospital visits on Physician reported global health burden | baseline to week 54
  Change in VAS on global health from 0 - 10 with higher values indicating a higher burden
Estimate effects of home monitoring compared to fixed-interval hospital visits on the disease activity in patients with rheumatoid arthritis associated ILD (RA-ILD) | baseline to week 54
  Change in Disease Activity Score-28 (DAS28)
Estimate effects of home monitoring compared to fixed-interval hospital visits on the disease activity in patients with Sjøgrens disease associated ILD (SjD-ILD) | baseline to week 54
  Change in EULAR Sjögren's syndrome disease activity index (ESSDAI)
Estimate effects of home monitoring compared to fixed-interval hospital visits on the disease activity in patients with inflammatory idiopathic myopathies including antisynthetasis syndromes on a visual analogue scales | baseline to week 54
  Change in MDAAT / MYOACT (range 0-60) where higher values would indicate more disease activity
Estimate effects of home monitoring compared to fixed-interval hospital visits on the disease activity in patients with inflammatory idiopathic myopathies including antisynthetasis syndromes on a questionnaire based skale | baseline to week 54
  Change in MDAAT / MITAX (range 0-63) where higher values would indicate more disease activity
Estimate effects of home monitoring compared to fixed-interval hospital visits on the disease activity in patients with systemic sclerosis | baseline to week 54
  Change in Revised European Scleroderma Trials and Research Group Activity Index (EUSTAR-AI) (range 0-10) where higher values would indicate more disease activity
Estimate effects of home monitoring compared to fixed-interval hospital visits on change in DLCO | at week 54
  Absolute change from baseline in DLCO (SI)
  · Absolute change from baseline in DLCO (% predicted)
Assess effect of home monitoring compared to fixed-interval hospital visits on extent of pulmonary fibrosis on high resolution computed tomography (HRCT) | baseline to week 54
  Change in extent of fibrosis as percentage of total lung parenchyma on HRCT
Estimate effects of home monitoring compared to fixed-interval hospital visits on degree of patient reported disability that breathlessness poses on day-to-day activities | baseline to week 54
  Change in "Modified Medical Research Council Dyspnoea Scale" (mMRC) with a range of 0-4 where higher values indicate more disability
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported dyspnea | baseline to week 54
  Change on a visual analogue scale for dyspnea where higher values would indicate more symptoms
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported cough | baseline to week 54
  Change on a visual analogue scale for cough where higher values would indicate more symptoms
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient reported symptoms | baseline to week 54
  Change on a visual analogue scale for fatigue where higher values would indicate more symptoms
Estimate ability of home monitoring compared to fixed-interval hospital visits to detect afebrile episodes | at week 54
  Number of verified afebrile episodes
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient treatment satisfaction | at week 54
  Difference in "Client satisfaction questionnaire 8" (CSQ-8) scores (range 8-32 where higher values indicate a higher satisfaction) between the to arms
Estimate effects of home monitoring compared to fixed-interval hospital visits on patient mental health parameters | at week 54
  Difference on the "Hosital Anxiety and Depression Scale" (HADS) with a range of 0-21 where higher scores would indicate more depression and axiety
Estimate the effects of home monitoring compared to fixed-interval hospital visits on identification of clinically significant Respiratory Tract Infections (csRTI) | at week 54
  Total number and proportion of severe csRTIs compared between the arms
Estimate the effects of home monitoring compared to fixed-interval hospital visits on length of antibiotic treatment due to clinically significant Respiratory Tract Infections (csRTI) | at week 54
  Days on antibiotic therapy for csRTIs compared between the arms
Estimate the effects of home monitoring compared to fixed-interval hospital visits on hospitalisation for clinically significant Respiratory Tract Infections (csRTI) | at week 54
  Days hospitalised for csRTIs compared between the arms
Estimate effects of home monitoring compared to fixed-interval hospital visits on identification of acute exacerbations | baseline to week 54
  Time to first acute exacerbation event
Assess immunologic activity in the peripheral blood by immune cells and soluble markers of inflammation in patients followed with home monitoring or fixed-interval hospital visits | at baseline and at week 54
  Assess content and change in peripheral blood markers derived from peripheral blood (as evaluated by sequencing techniques, proteomics and cellular phenotyping)
Assess immunologic activity in nasal swabs by immune cells and soluble markers of inflammation in patients followed with home monitoring or fixed-interval hospital visits | at baseline and at week 54
  Assess content and change in immune cells and soluble markers of inflammation in nasal swabs (as evaluated by sequencing techniques, proteomics and cellular phenotyping)
Estimate effects of home monitoring compared to fixed-interval hospital visits on changes in immunosuppressive therapy | baseline to week 54
  Proportion of participants subjected to increased immunosuppression
Assess remission of non-ILD disease manifestations in patients followed with home monitoring or fixed-interval hospital visits | at baseline and at week 54
  Proportion of participants in non-remission for non-ILD disease manifestations
Assess the effect of reflux disease at baseline on ILD progression | after 54 weeks
  Proportion of patients who experience ILD progression with reflux disease compared to no reflux disease

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Maria Hoffmann-Vold, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
The individual patient data of this study will not be publicly available as they contain information that could compromise the privacy of research participants and may be subject to ongoing research as long as the research project is ongoing. The original data will be available from the corresponding authors of subsequent publications upon reasonable request, except where restricted by GDPR liabilities.

REFERENCES:
- See also: University homepage — https://www.oslo-universitetssykehus.no/avdelinger/Klinikk-for-kirurgi-og-spesialisert-medisin/avdeling-for-revmatologi-hud-og-infeksjonssykdommer/seksjon-for-revmatologi/forskningsprosjekter/nor-milder/